CLINICAL TRIAL: NCT02395991
Title: Evaluation of Transient Dyspnea During Gadoxetic Acid Enhanced Multiphasic Liver MRI
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, MD, Seoul National University Hospital
Other Study IDs: CS_2015_ISS
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Dyspnea
Keywords: gadoxetic acid; transient dyspnea
MeSH Terms: conditions — Dyspnea | interventions — gadolinium ethoxybenzyl DTPA; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observe1: Patients who are referred to MR unit for hepatocyte-specific contrast (gadoxetic acid) enhanced liver magnetic resonance imaging (MRI)
  Interventions: Drug: gadoxetic acid; Other: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Drug: gadoxetic acid — standard dose of gadoxetic acid (0.025mmol/kg) intravenous administration
  Other Names: eovist; primovist
Other: Magnetic resonance imaging (MRI) — Dynamic T1 weighted sequence consist of precontrast, arterial, portal, transitional and hepatobiliary phases.
  precontrast, arterial and portal phases (prior to contrast media injection to 60 seconds after contrast media injection) are obtained continuously in free-breathing state. Transitional and hepatobiliary phases are obtained in breath-hold state.

SUMMARY:
The purpose of this study is to observe transient dyspnea pattern after Gd-EOB-DTPA administration by obtaining continuous dynamic T1 weighted image data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred to MR unit for hepatocyte-specific contrast enhanced liver MRI using gadoxetic acid, to characterize focal liver lesion or to investigate diffuse liver disease
* OR, Liver living donor candidates
* AND subjects who sign the informed consent.

Exclusion Criteria:

* Minors under 18 years old
* All contraindication to MRI
* Hypersensitivity to Gd
* Biliary obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred to MR unit for hepatocyte-specific contrast enhanced liver MRI using gadoxetic acid.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2015 to October 2015, patients who are referred to Radiology unit in SNUH for liver MRI scan.
Groups:
- EOB-MRI: Patients who are referred to MR unit for hepatocyte-specific contrast (gadoxetic acid) enhanced liver magnetic resonance imaging (MRI)
  gadoxetic acid: standard dose of gadoxetic acid (0.025mmol/kg) intravenous administration
  Magnetic resonance imaging (MRI): Dynamic T1 weighted sequence consist of precontrast, arterial, portal, transitional and hepatobiliary phases.
  precontrast, arterial and portal phases (prior to contrast media injection to 60 seconds after contrast media injection) are obtained continuously in free-breathing state. Transitional and hepatobiliary phases are obtained in breath-hold state.
Period: Overall Study
Arm/Group | EOB-MRI
Started | 60
Completed | 59
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Observe1: Patients who are referred to MR unit for hepatocyte-specific contrast (gadoxetic acid) enhanced liver magnetic resonance imaging (MRI)
  gadoxetic acid: standard dose of gadoxetic acid (0.025mmol/kg) intravenous administration
  Magnetic resonance imaging (MRI): Dynamic T1 weighted sequence consist of precontrast, arterial, portal, transitional and hepatobiliary phases.
  precontrast, arterial and portal phases (prior to contrast media injection to 60 seconds after contrast media injection) are obtained continuously in free-breathing state. Transitional and hepatobiliary phases are obtained in breath-hold state.
Arm/Group | Observe1
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35
Region of Enrollment [Number; unit: participants]
  South Korea | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Transient Dyspnea.
Description: A sudden onset irregular breathing pattern after EOB administration, based on MRI k-space data (not participants' symptom).
  The k-space data was analyzed after the enrollment completion.
Time Frame: during 3 minutes after contrast media administration
Measure: Count of Participants; unit: Participants
Arm/Group | EOB-MRI
Number analyzed (Participants) | 59
Participants | 23

2. Secondary Outcome: Duration of Transient Dyspnea in Participants With Transient Dyspnea.
Description: The duration of transient dyspnea was analyzed based on the MRI k-space data, using a dedicated software.
  The analysis using the MRI k-space data was performed after the completion of enrollment.
Time Frame: during 3 minutes after contrast media administration
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Observe1
Number analyzed (Participants) | 59
second | 21.5 (13)

3. Other Pre Specified Outcome: Liver Stiffness Value
Description: liver stiffness value from MR elastography using GRE and SE sequence which is a part of protocol.
  Both GRE and SE sequences are two different sequences for obtaining MR elastogrphy which measures the stiffness of the liver.
  The measured liver stiffness is known to be related to the degree of hepatic fibrosis and/or inflammation.
Time Frame: in three days after MRI
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | EOB-MRI
Number analyzed (Participants) | 59
kPa
  SE MRE | 3.87 (1.19)
  GRE MRE | 3.76 (1.29)

ADVERSE EVENTS:
Time Frame: 1 hour after MRI completion
Arm/Group | EOB-MRI
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes